CLINICAL TRIAL: NCT05601323
Title: A Randomized Controlled Study of Suizenji in Patients With Unresectable Pancreatic Cancer
Brief Title: A Study of Suizenji in Patients With Unresectable Pancreatic Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: SONIRE Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Sonire-PAC-001
Record Dates: First submitted 2022-10-27; First posted 2022-11-01 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Unresectable Pancreatic Cancer
Keywords: Unresectable Pancreatic Cancer; Suizenji; high intensity focused ultrasound; HIFU

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- HIFU (High-Intensity Focused Ultrasound) + Chemotherapy (Experimental): HIFU treatment with Suizenji: up to 2 times per week (1 course) for pancreatic primary lesions; the second course should be at least 60 days apart, up to a maximum of 5 courses.
  Chemotherapy (physician's choice): Nal-IRI/FL, mFOLFIRINOX or Gem/nab-PTX
  Interventions: Device: Suizenji; Drug: Nal-IRI/FL; Drug: mFOLFIRINOX; Drug: Gem/nab-PTX
- Chemotherapy (Active Comparator): Chemotherapy (physician's choice): Nal-IRI/FL, mFOLFIRINOX or Gem/nab-PTX
  Interventions: Drug: Nal-IRI/FL; Drug: mFOLFIRINOX; Drug: Gem/nab-PTX

INTERVENTIONS:
Device: Suizenji — HIFU treatment
  Arms: HIFU (High-Intensity Focused Ultrasound) + Chemotherapy
Drug: Nal-IRI/FL — Nanoliposomal irinotecan, Fluorouracil, Levofolinate
Drug: mFOLFIRINOX — Fluorouracil, Levofolinate, Irinotecan, Oxaliplatin
Drug: Gem/nab-PTX — Gemcitabine, nab-Paclitaxel

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of standard chemotherapy with or without a novel High Intensity Focused Ultrasound system (Code: Suizenji) in patients with unresectable pancreatic cancer who are refractory or intolerant to first-line chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Ages 20 years and over.
* Unresectable pancreatic cancer (including metastatic pancreatic cancer) who are refractory or intolerant to first-line chemotherapy. Any first-line chemotherapy is acceptable.
* Target treatment tumor is located in the pancreas, and the target tumor can be visualized with ultrasound echography and can also be treated by high-intensity focused ultrasound.
* Has primary tumor site of measurable lesion according to RECIST guidelines version 1.1
* ECOG performance status of 0 to 2.

Exclusion Criteria:

* Active multiple cancers that require treatment.
* Suspected gastrointestinal invasion of the primary tumor based on CT scan.
* Obstructive jaundice. However, patients who have a bile duct stent placed for obstructive jaundice by the time of allocation may be enrolled.
* Child-Pugh Classification B or C liver failure due to liver metastases.
* Tumor embolization in the veins surrounding the pancreas.
* Cystic component within the pancreatic cancer.
* Peritoneal dissemination.
* Pleural effusion or ascites with poorly controlled
* Contraindications to the use of secondary chemotherapy used in this study.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-01-31 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | Up to approximately 24 months

SECONDARY OUTCOMES:
Progression-free survival | Up to approximately 12 months
1-year survival rate | Up to approximately 12 months
Objective response rate | Up to approximately 12 months
Disease control rate | Up to approximately 12 months
Adverse Events | Up to approximately 12 months

CONTACTS AND LOCATIONS:
Overall Officials: SONIRE Therapeutics Inc., Study Director — SONIRE Therapeutics Inc.
Locations (7):
- Japan (7):
  - Aichi Medical University Hospital, Nagakute-shi, Aichi
  - Tohoku University Hospital, Sendai-shi, Miyagi
  - Tokyo Medical University Hospita, Shinjuku-ku, Tokyo
  - Toyama University Hospital, Toyama-shi, Toyama
  - Wakayama Medical University Hospital, Wakayama-shi, Wakayama
  - Yokohama City University Medical Center, Yokohama-shi, Kanagawa
  - Kanagawa Cancer Center, Yokohama-shi, Kanagawa

IPD SHARING:
Plan to Share IPD: No